CLINICAL TRIAL: NCT04884646
Title: Effects of Virtual Reality Versus Motor Imagery Versus Routine Physical Therapy in Patients With Parkinson's Disease: A Randomised Controlled Trial
Brief Title: Effects of Virtual Reality Versus Motor Imagery Versus Routine Physical Therapy in Patients With Parkinson's Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Fsd/0115
Record Dates: First submitted 2021-05-07; First posted 2021-05-13 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Parkinson Disease
Keywords: Parkinson; Virtual Reality; Motor Imagery; Routine Physical Therapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study would be single blinded as accessor of the study would be kept blind of the treatment group to which patient would be allocated.After the complete initial screening process, every recruited patient will be accessed by an independent assessor, expert will use outcome measuring tools. his will be recorded as baseline measurement assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality with Routine Physical Therapy (Experimental): The duration of the VR will be from 10 to 15 minutes during each session and Routine Physical Therapy for 40 minutes which consists of warming-up, stretching, strengthening and active exercises for relaxation, coordination exercises for limbs, trunk, neck, and gait training)
  Interventions: Other: VR with Routine physical therapy and Virtual reality
- Motor imagery technique with Routine Physical Therapy (Experimental): Motor Imagery techniques will be given for 5 to 10 minutes along with routine physical therapy for 40 minutes which consists of warming-up, stretching, strengthening and active exercises for relaxation, coordination exercises for limbs, trunk, neck, and gait training)
  Interventions: Other: Motor Imagery with Routine physical therapy
- Routine Physical Therapy (Experimental): Only routine physical therapy will be given (including warming-up, stretching, strengthening and active exercises for relaxation, coordination exercises for limbs, trunk, neck, and gait training)
  Interventions: Other: Routine physical therapy

INTERVENTIONS:
Other: VR with Routine physical therapy and Virtual reality — VR group will be treated with virtual reality for 15 to 20 minutes along with routine physical therapy for 40 minutes session 3 days/week for 12 weeks
  Other Names: Rehabilitation following VR with Routine physical therapy treatment
  Arms: Virtual Reality with Routine Physical Therapy
Other: Motor Imagery with Routine physical therapy — MI group will be treated with virtual reality for 15 to 20 minutes along with routine physical therapy for 40 minutes session 3 days/week for 12 weeks
  Other Names: Rehabilitation following MI with Routine physical therapy treatment
  Arms: Motor imagery technique with Routine Physical Therapy
Other: Routine physical therapy — Group A will be given routine physical therapy in 40-min sessions and 20 min of walking and cycling with a short period of rest, every alternate day (3 days per week) for 12 weeks
  Other Names: Rehabilitation following Routine physical therapy treatment
  Arms: Routine Physical Therapy

SUMMARY:
The aim of this study is to investigate the effects of VR and MI techniques in addition to routine physical therapy on motor skills, balance and ADL in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease is one of the most common, insidious neurological disorders with major motor symptoms, including bradykinesia, resting tremors, rigidity, and postural disorders. Virtual reality and motor imagery are among the more innovative techniques for rehabilitation of patients with Parkinson's disease that promote motor learning through both explicit and implicit processes.This study is unique in that it examines the effects of VR versus MI on motor skills, balance, and daily living activities in individuals with Parkinson's disease

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease
* Modified Hoehn and Yahr Scale(H&Y stages I to III)
* Between the ages of 50 and 80 years of both genders
* Independent in transfers
* A score equal to or greater than 24 on the Mini-Mental State Examination (MMSE), and
* Previous lack of participation in balance or motor training.

Exclusion Criteria:

* History of any neurological conditions such as stroke, multiple sclerosis, epilepsy other than Parkinson's disease,
* History of orthopedic issues such as pain, fracture, or lower limb pathology,
* History of visual abnormalities,
* History of any chronic or cardiovascular pathology that can interfere with the transfer procedure or can affect the training sessions,
* The participants having severe dyskinesia or "on-off" phases,
* Previous history of surgery for PD,
* History of virtual games used for treatment in the past three months, and
* Virtual game phobia.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2021-06-12 (Actual)

PRIMARY OUTCOMES:
Unified Parkinson's disease Rating Scale Part II | 3 months
  This is a subjective instrument that is widely used in clinical settings for patients with Parkinson's disease. This scale comprises 31 elements, which are divided into three sub-scales: Sub-scale II comprises the evaluation of activities in daily living. A possible maximum of 199 points can be scored on this scale. A score of 199 refers to complete disability and 0 refers to the absence of disability .
Unified Parkinson's disease Rating Scale Part III | 3 months
  This is a subjective instrument that is widely used in clinical settings for patients with Parkinson's disease. This scale comprises 31 elements, which are divided into three sub-scales and sub-scale III evaluates the motor system. A possible maximum of 199 points can be scored on this scale. A score of 199 refers to complete disability and 0 refers to the absence of disability
Berg Balance Scale (BBS) | 3 months
  The scale has been established as the most widely used assessment tool in clinical settings to identify changes in balance performance. A score of less than 45 is considered a limit for the risk of falling, while a score of 56 relates to functional balance

SECONDARY OUTCOMES:
Activities-specific Balance Confidence Scale (ABC): | 3 months
  This scale is used as a predictor of falls in patients with neurological deficits. Patients are rated from 0% to 100%, with 0% interpreted as not at all safe and 100% as completely safe

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No